CLINICAL TRIAL: NCT01297504
Title: A One-Year Observational Study of Palivizumab in Infants at Risk for Respiratory Syncytial Virus Infection in Latin America
Brief Title: A One-Year Observation of Palivizumab in Infants at Risk for Respiratory Syncytial Virus Infection in Latin America
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Fundasamin (Argentina) (Unknown)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-129
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: palivizumab; lower respiratory tract infection; Respiratory syncytial virus; usage patterns
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Palivizumab: Infants at risk for respiratory syncytial virus infection received palivizumab prescribed in accordance with the terms of the local marketing authorization.

SUMMARY:
The study was designed to gather information regarding the use of palivizumab for the prophylaxis for respiratory syncytial virus (RSV) infection in high-risk infants in selected countries within Latin America.

DETAILED DESCRIPTION:
RSV causes significant disease. There is a paucity of data from developing countries even though existing data clearly indicate that RSV accounts for a high proportion of acute respiratory illnesses (ARIs) in children.

This is a multi-center study in a cohort of infants at risk for RSV infection in Latin America who have received palivizumab in the usual manner in accordance with the terms of marketing authorization with regard to dose, population and indication. Enrolled participants were followed for one year after their first dose of palivizumab. Epidemiological and clinical data as well as information about compliance, hospitalizations and safety was collected.

ELIGIBILITY:
Inclusion Criteria:

* Children with a history of bronchopulmonary dysplasia, infants with a history of prematurity (less than or equal to 35 weeks gestational age), or children with hemodynamically significant congenital heart disease who received the first dose of palivizumab within the 2 weeks prior to the signature of the Informed Consent Form.
* Parent or legal guardian of child provides written Informed Consent

Exclusion Criteria:

* Children excluded from receiving palivizumab as per local guidelines

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study was conducted at primary care clinics in Latin America.
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2011-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Castillo, MD, Study Director — Abbvie S.A.
Locations (24):
- Argentina (4):
  - Site Reference ID/Investigator# 52185, Buenos Aires
  - Site Reference ID/Investigator# 52182, Buenos Aires
  - Site Reference ID/Investigator# 52183, Buenos Aires
  - Site Reference ID/Investigator# 52184, Buenos Aires
- Chile (2):
  - Site Reference ID/Investigator# 54426, Santiago
  - Site Reference ID/Investigator# 54427, Santiago
- Colombia (10):
  - Site Reference ID/Investigator# 52732, Armenia
  - Site Reference ID/Investigator# 52722, Barranquilla
  - Site Reference ID/Investigator# 52726, Barranquilla
  - Site Reference ID/Investigator# 52723, Bogotá
  - Site Reference ID/Investigator# 52725, Bogotá
  - Site Reference ID/Investigator# 52727, Bogotá
  - Site Reference ID/Investigator# 52729, Bogotá
  - Site Reference ID/Investigator# 63882, Bogotá
  - Site Reference ID/Investigator# 52735, Cali
  - Site Reference ID/Investigator# 52731, Medellín
- Ecuador (2):
  - Site Reference ID/Investigator# 52703, Quito
  - Site Reference ID/Investigator# 52704, Quito
- Mexico (3):
  - Site Reference ID/Investigator# 52082, Guanajuato, Leon
  - Site Reference ID/Investigator# 52084, Mexico City, DF
  - Site Reference ID/Investigator# 52083, Nuevo Leon, Monterrey
- Peru (2):
  - Site Reference ID/Investigator# 52243, Callao
  - Site Reference ID/Investigator# 52242, Lima
- Site Reference ID/Investigator# 52246, Salto, Uruguay

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palivizumab
Started | 464
Participants Studied | 458 (Six participants were eliminated due to invalid consent, previous palivizumab or no study visits)
Completed | 397
Not Completed | 67
Not completed — Invalid Consent | 1
Not completed — Received Palivizumab in Previous Season | 1
Not completed — No Study Visits | 4
Not completed — Death | 3
Not completed — Lost to Follow-up | 43
Not completed — Withdrawal by Subject | 9
Not completed — Site Closure | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: Participants Studied
Arm/Group | Palivizumab
Number analyzed (Participants) | 458
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 55 [31 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219
  Male | 239
Region of Enrollment [Number; unit: participants]
  Mexico | 100
  Ecuador | 7
  Argentina | 149
  Uruguay | 10
  Peru | 13
  Chile | 32
  Colombia | 147
Birth Weight [Mean (Standard Deviation); unit: g] | 1344.6 (460.5)

OUTCOME MEASURES:

1. Primary Outcome: Characterization of Participants With Risk Factors for Respiratory Syncytial Virus (RSV) Infection
Description: Study participants were characterized at Baseline by history of bronchopulmonary dysplasia, history of prematurity (less than or equal to 35 weeks gestational age), children with hemodynamically significant congenital heart disease (CHD), the presence of cohabitants less than 6 years old, possible exposure to indoor tobacco smoke, day care attendance, asthmatic or atopic mother, smoking during pregnancy, breastfeeding, prenatal assistance (4 or more visits during pregnancy), neonatal hospitalization care, history of neonatal assisted ventilation, and mother education level (completed primary school).
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 458
participants
  History of bronchopulmonary dysplasia | 134
  Prematurity | 449
  Congenital heart disease | 46
  Presence of cohabitants <6 years of age | 160
  Smoking at home | 78
  Day care attendance | 5
  Asthmatic / atopic mother | 55
  Smoking during pregnancy | 9
  Breastfeeding | 336
  Prenatal assistance | 386
  Neonatal care hospitalization | 447
  History of neonatal assisted ventilation | 257
  Mother education level | 443

2. Secondary Outcome: Number of Participants With Hospitalizations for Lower Respiratory Tract Infection and RSV
Description: The number of participants with hospitalizations due to lower respiratory tract infection (LRTI) and hospitalizations due to lower respiratory tract infection caused by RSV.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 458
participants
  Hospitalization due to LRTI | 52
  Hospitalization due to LRTI due to RSV | 12

3. Secondary Outcome: Characterization of Hospitalization Episodes Due to Lower Respiratory Tract Infection and RSV
Time Frame: 12 months
Population: Participants with hospitalization due to LTRI and hospitalization due to LTRI and RSV.
Measure: Number; unit: hospitalization episodes
Units Other Than Participants: Hospitalization episodes
Groups:
- LTRI: Hospitalizations due to lower respiratory tract infections (LRTI).
- LTRI Due to RSV: Hospitalizations due to lower respiratory tract infections (LRTI) caused by RSV
Arm/Group | LTRI | LTRI Due to RSV
Number analyzed (Participants) | 52 | 12
Number analyzed (Hospitalization episodes) | 61 | 12
hospitalization episodes
  Prematurity | 60 | 12
  Bronchopulmonary dysplasia | 32 | 9
  Congenital heart disease | 7 | 1

4. Secondary Outcome: Risk Factors for Hospitalization
Description: Variables that could act as risk factors for hospitalization for lower respiratory tract infection were tested in univariate and multivariate Poisson regression models. Baseline characteristics, such as age, gender, birth weight and comorbidities were included as covariates in the Poisson regression model. Variables for multivariate analysis were added applying forward selection. Gestational age and birth weight were included as continuous variables, considering that the higher they were the better they could act as a protection factor for hospitalization due to respiratory infection.
Time Frame: Baseline and 12 months
Measure: Number (95% Confidence Interval); unit: rate ratio
Arm/Group | Univariate | Multivariate
Number analyzed (Participants) | 458 | 458
rate ratio
  Sex (Female) | 0.919 [0.553 to 1.528] | 0.925 [0.545 to 1.569]
  Gestational Age | 0.925 [0.84 to 1.018] | 1.022 [0.866 to 1.207]
  Bronchopulmonar Dysplasia | 2.768 [1.667 to 4.597] | 2.754 [1.53 to 4.957]
  Cardiopathy | 1.149 [0.494 to 2.671] | 0.925 [0.378 to 2.265]
  Smoking | 2.546 [0.797 to 8.130] | 1.36 [0.378 to 4.889]
  Birth Weight | 0.9996 [0.9989 to 1.0002] | 0.9998 [0.999 to 1.001]
  Compliance | 1.004 [0.995 to 1.013] | 1.005 [0.996 to 1.014]
  Maternal Education (elementary) | 2.108 [1.038 to 4.282] | 1.84 [0.849 to 3.989]

5. Secondary Outcome: Compliance to Prescribed Palivizumab
Description: Compliance to prescribed palivizumab was calculated based on the number of doses received versus the expected number of doses for each participant. The expected number of doses for each participant was estimated based on seasonality and current prescription guidelines for each country.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of expected dose
Arm/Group | Palivizumab
Number analyzed (Participants) | 458
Percentage of expected dose | 83.66 [80.83 to 86.48]

6. Primary Outcome: Distribution of Comorbidities in Study Participants
Description: The percentage of participants with each and combinations of the three comorbidities for which palivizumab is indicated.
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 458
percentage of participants
  Prematurity only | 64.63
  Bronchopulmonary dysplasia (BPD) only | 0.87
  Congenital heart disease (CHD) only | 0.87
  BPD + Prematurity | 24.45
  Prematurity + CHD | 5.24
  Prematurity + BPD + CHD | 3.71
  BPD + CHD | 0.22

7. Secondary Outcome: Mean Number of Doses of Palivizumab Administered
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Palivizumab
Number analyzed (Participants) | 458
doses | 3.8 (1.26)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Palivizumab
Serious Adverse Events (participants affected / at risk) | 102/458
Other Adverse Events (participants affected / at risk) | 299/458
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab (N=458)
Acute prerenal failure (Renal and urinary disorders) | 1
Apparent life-threatening event (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1
Infantile apneic attack (Respiratory, thoracic and mediastinal disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 16
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5
Bacterial infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 3
Bronchiolitis (Infections and infestations) | 28
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenterocolitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 6
Haemophilus infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Lung infection pseudomonal (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Obstructive bronchitis (Infections and infestations) | 1
Otitis media recurrent (Infections and infestations) | 1
Parainfluenzae viral laryngotracheobronchitis (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 8
Pneumonia bacterial (Infections and infestations) | 3
Pneumonia chlamydial (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 7
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Sepsis neonatal (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 3
Convulsion (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Infantile spasms (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Milk allergy (Immune system disorders) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Gastrointestinal atoma complication (Injury, poisoning and procedural complications) | 1
Retinopathy of prematurity (Eye disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 11
Jugular vein thrombosis (Vascular disorders) | 1
Haemodynamic instability (Vascular disorders) | 1
Heart failure (Cardiac disorders) | 1
Pallor (Vascular disorders) | 2
Subvalvular aortic stenosis (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal mass (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 9
Gastroesophageal reflux disease (Gastrointestinal disorders) | 11
Haematochezia (Gastrointestinal disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 5
Meconium ileus (Gastrointestinal disorders) | 1
Megacolon (Gastrointestinal disorders) | 1
Reflux gastritis (Gastrointestinal disorders) | 1
Stools watery (Gastrointestinal disorders) | 1
Volvulus of small bowel (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 11
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 1
Feeding disorder (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Food intolerance (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 3
Malnutrition (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1
Underweight (Metabolism and nutrition disorders) | 1
Weight gain poor (Metabolism and nutrition disorders) | 1
Death (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Hyperthermia (General disorders) | 1
Pyrexia (General disorders) | 18
Malaise (General disorders) | 3
Mucosal Inflammation (General disorders) | 1
Irritability (General disorders) | 3
General physical health deterioration (General disorders) | 2
Arterial septal defect (Congenital, familial and genetic disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Atrioventricular septal defect (Congenital, familial and genetic disorders) | 1
Intestinal malrotation (Congenital, familial and genetic disorders) | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1
Heart disease congenital (Congenital, familial and genetic disorders) | 1
Hypospadias (Congenital, familial and genetic disorders) | 2
Laryngomalacia (Congenital, familial and genetic disorders) | 1
Pilonidal cyst congenital (Congenital, familial and genetic disorders) | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Anaemia neonatal (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hepatoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CSF test abnormal (Investigations) | 1
Oxygen saturation decreased (Investigations) | 5
Oxygen consumption increased (Investigations) | 1
Respiratory syncytial virus test positive (Investigations) | 3
Urine analysis abnormal (Investigations) | 1
Urine output decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Agitation (Psychiatric disorders) | 1
Tracheostomy (Surgical and medical procedures) | 1
Inguinal hernia repair (Surgical and medical procedures) | 1
Oral surgery (Surgical and medical procedures) | 1
Ophthalmic fluid drainage (Surgical and medical procedures) | 1
Vascular operation (Surgical and medical procedures) | 1
Hypotonia neonatal (Musculoskeletal and connective tissue disorders) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 2
Feeding disorder neonatal (Metabolism and nutrition disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab (N=458)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 73
Diarrhoea (Gastrointestinal disorders) | 52
Pyrexia (General disorders) | 49
Bronchiolitis (Infections and infestations) | 71
Ear infection (Infections and infestations) | 23
Dermatitis (Skin and subcutaneous tissue disorders) | 23
Rash (Skin and subcutaneous tissue disorders) | 23
Upper respiratory tract infection (Infections and infestations) | 242

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.